CLINICAL TRIAL: NCT01535898
Title: Application of High Resolution Diffusion-weighted MR Imaging Pulse Sequence in Head and Neck, and Prostate Cancers
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 12-033
Record Dates: First submitted 2012-02-13; First posted 2012-02-20 (Estimated); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: Head and Neck Cancer; Prostate Cancer
Keywords: MRI; MR imaging Pulse Sequence; High Resolution Diffusion-weighted; Questionnaire; 12-033
MeSH Terms: conditions — Head and Neck Neoplasms; Prostatic Neoplasms | interventions — Base Sequence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Pts having an MRI: This is a technology assessment protocol. The study is designed to assess the utility of the technology using a limited number of participants.
  Interventions: Other: MRI scanner with sequence

INTERVENTIONS:
Other: MRI scanner with sequence — The intervention for the patients is the additional 10 minutes in the MRI scanner with sequence. The intervention for the volunteers is the scan, which will take a total of 30 minutes. The volunteers will have two more additional studies at 1-2 week intervals. Both the patients and volunteers will also need to fill out a questionnaire.

SUMMARY:
Magnetic resonance imaging (MRI) is a diagnostic study that makes pictures of organs of the body using magnetic field and radio frequency pulses that can not be felt. The purpose of this study is to determine if a new MR imaging method can help tumor evaluation in head and neck cancer or prostate cancer. The extra images will be obtained using Diffusion-weighted Magnetic Resonance Imaging which provides image contrast through detection of small restrictions in the movement of water molecules. This study may help us provide additional information about the tumor along with the picture of the organ.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 and over.
* Men and women without regard to ethnic background.
* Patients/Subjects able to give informed consent
* Patients/Subjects whose weight does not exceed 275 lbs.
* Patient with a known or suspected head and neck cancer or prostate cancer scheduled for an MRI scan as part of their routine care --OR--
* Volunteer with no history of the disease in that category.

Exclusion Criteria:

* Patients who are unwilling or unable to undergo MRI including patients with contra-indications to MRI such as the presence of cardiac pacemakers or non-compatible intracranial vascular clips.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The radiologists on the study will identify potential research participants from those patients who are scheduled for MRI examination as part of their routine clinical care.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2012-02; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
feasibility of high resolution diffusion-weighted imaging | 2 years
  using a new DWI pulse sequence from the manufacturer (General Electric Medical Systems (Milwaukee, WI)) for the assessment of head and neck cancer cancer and prostate cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Amita Dave, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/